CLINICAL TRIAL: NCT03872778
Title: A Phase I/IIa Open-label, Multi-center Study to Evaluate the Safety, Tolerabiity, Whole-body Distribution, Radiation Dosimetry and Anti-tumor Activity of [177Lu]-NeoB Administered in Patients With Advanced Solid Tumors Known to Overexpress Gastrin-releasing Peptide Receptor (GRPR)
Brief Title: [177Lu]-NeoB in Patients With Advanced Solid Tumors and With [68Ga]-neoB Lesion Uptake
Acronym: NeoRay
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAAA603A12101; 2023-507170-41-00 (Registry Identifier: EU CTIS number)
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms
Keywords: AAA603; [177Lu]-NeoB; [68Ga]-neoB; whole-body distribution; radiation dosimetry; anti-tumor activity; Advanced solid tumors; Overexpress gastrin-releasing peptide receptor; GRPR; Lutetium-177 (177Lu)
MeSH Terms: conditions — Neoplasms | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Intervention Model Description: Phase I: dose range finding to identify Recommended Phase II Dose Phase IIa: assessment of anti-tumor activity
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Phase I Cohort 1 (DL1(50mCi + 150mCi) (Experimental): Participants received the 1.85 GBq (50mCi) +/- 10% of [177Lu]-NeoB at cycle 1 and then received 5.55 GBq (150mCi）+/- 10% of [177Lu]-NeoB for at least 3 cycles.
  Interventions: Drug: [177Lu]-NeoB; Drug: [68Ga]-NeoB
- Phase I Cohort 2 (DL2 200mCi) (Experimental): Participants received the 9.25 GBq (250mCi) +/- 10% of [177Lu]-NeoB once every 6 weeks for at least 3 cycles.
  Interventions: Drug: [177Lu]-NeoB; Drug: [68Ga]-NeoB
- Phase I Cohort 3 (DL3 250mCi) (Experimental): Participants received the 11.1 GBq (300mCi) +/- 10% of [177Lu]-NeoB once every 6 weeks for at least 3 cycles.
  Interventions: Drug: [177Lu]-NeoB; Drug: [68Ga]-NeoB
- Phase II Cohort A (Breast Cancer) (Experimental): Participants received the 9.25 GBq (250mCi) +/- 10% of [177Lu]-NeoB once every 6 weeks for at least 3 cycles.
  Interventions: Drug: [177Lu]-NeoB; Drug: [68Ga]-NeoB
- Phase II Cohort B (Prostate Cancer) (Experimental): Participants received the 9.25 GBq (250mCi) +/- 10% of [177Lu]-NeoB once every 6 weeks for at least 3 cycles.
  Interventions: Drug: [177Lu]-NeoB; Drug: [68Ga]-NeoB
- Phase II Cohort C (Gastro Intestinal Stromal Tumor (GIST)) (Experimental): Participants received the 9.25 GBq (250mCi) +/- 10% of [177Lu]-NeoB once every 6 weeks for at least 3 cycles.
  Interventions: Drug: [177Lu]-NeoB; Drug: [68Ga]-NeoB
- Phase II Cohort D (Renal Impairment) (Experimental): These were participants with any advanced/metastatic solid tumor type, and with moderate impaired renal function. The participants received the 9.25 GBq (250mCi) +/- 10% of [177Lu]-NeoB once every 6 weeks for at least 3 cycles.
  Interventions: Drug: [177Lu]-NeoB; Drug: [68Ga]-NeoB
- Phase II Cohort E (Breast, Prostate, GIST) (Experimental): These participants were eligible for enrollment in any of the three advanced/metastatic tumor type (as defined for cohorts A,B,C. The participants received the 5.55 GBq (150mCi) +/- 10% of [177Lu]-NeoB and neprilysin inhibitor (NEPi) LCZ696 in cycle 1 and then 9.25 GBq (250mCi) +/- 10% of [177Lu]-NeoB once every 6 weeks for at least 3 cycles.
  Interventions: Drug: [177Lu]-NeoB; Drug: [68Ga]-NeoB; Drug: LCZ696

INTERVENTIONS:
Drug: [177Lu]-NeoB — [177Lu]-NeoB: peptide receptor radionuclide therapy
  Other Names: Lutetium NeoB, AAA603
Drug: [68Ga]-NeoB — [68Ga]-NeoB radioactive diagnostic agent
  Other Names: Gallium NeoB
Drug: LCZ696 — dose strength 49/51 mg, film-coated tablets for oral use
  Other Names: sacubitril/valsartan
  Arms: Phase II Cohort E (Breast, Prostate, GIST)

SUMMARY:
First in Human (FIH) study to characterize the safety, tolerability, pharmacokinetics (PK), distribution, radiation dosimetry, and anti-tumor activity of [177Lu]-NeoB in patients with advanced solid tumors known to overexpress GRPR and with [68Ga]-NeoB lesion uptake.

DETAILED DESCRIPTION:
This study was designed to establish whether the ligand NeoB, a high affinity antagonist for GRPR, could be used in a theragnostic approach for selection and therapy of GRPRexpressing malignancies: radiolabeled with (1) Gallium 68 (68Ga) to identify lesions and with (2) Lutetium-177 (177Lu) for the treatment of these lesions.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to participation
* Adult patients with advanced solid tumors known to overexpress GRPR
* [68Ga]-NeoB tumor lesion uptake on PET/CT or PET/MRI scan at screening visit (>50% of lesions detected with conventional imaging are identified as well by [68Ga]-NeoB uptake)
* At least one measurable lesion per RECIST 1.1/RANO with a [68Ga]-NeoB uptake
* Patients for whom no standard therapy is available, tolerated or appropriate
* Presence of at least one tumor lesion confirmed with functional or structural imaging (PET, SPECT, CT, MRI, bone scan) within 2 months prior to study entry
* Patient Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Life expectancy more than 6 months.

Exclusion Criteria:

* Creatinine clearance (calculated using Cockcroft-Gault formula, or measured) < 60 mL/min or serum creatinine > 1.5 x ULN.
* Platelet count of < 75 x 10e9/L
* Absolute neutrophil count (ANC) < 1.0 x 10e9/L
* Hemoglobin < 9 g/dL
* alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 x upper limit of normal (ULN) if no demonstrable liver metastases of > 5 x ULN in the presence of liver metastases
* Total bilirubin > 1.5 ULN, except for patients with documented Gilbert's syndrome who are eligible if total bilirubin ≤ x ULN
* Serum amylase and/or lipase > 1.5 ULN
* Known or expected hypersensitivity to [177Lu]-NeoB, [68Ga]-NeoB or any of their excipients
* Impaired cardiac function or clinically significant cardiac disease, including any of the following:

  * Clinically significant and/or uncontrolled heart disease such as congestive heart failure requiring treatment (New York Heart Association (NHYA) grade ≥2), uncontrolled arterial hypertension or clinically significant arrhythmia
  * LVEF < 50% as determined by echocardiogram (ECHO)
  * QTcF > 470 msec for females and QTcF >450 msec for males on screening electrocardiogram (ECG) or congenital long QT syndrome
  * Acute myocardial infarction or unstable angina pectoris < 3 months prior to study entry
* Patients with diabetes mellitus requiring insulin treatment and/or with clinical signs or with fasting plasma glucose > 160 mg/dL (8.9 mmol/L)
* Patients with history of or ongoing acute or chronic pancreatitis
* Prior administration of a radiopharmaceutical with therapeutic intent within a period corresponding to 10 half-lives of the radionuclide used in such radiopharmaceutical
* Prior External Beam Radiation Therapy (EBRT) to more than 25% of the bone marrow
* Patients with a bone scan showing an excessive skeletal radiopharmaceutical uptake with absent or faint activity in soft tissues and the genitourinary tract due to diffuse bone/bone marrow metastases in bone scan also called a "superscan"
* Prior treatment with Radium=223
* Patients who have changed the dose of systemic steroid therapy within less than 2 weeks prior to study entry or patients for whom steroid dose increase is anticipated during the study.
* Patients who have received prior systemic anti-cancer treatment within the following time frames:

  * Cyclical chemotherapy within a period that is shorter than the cycle length used for that treatment (e.g. 6 weeks for nitrosourea, mitomycin-C) prior to starting study treatment
  * Biologic therapy (e.g. antibodies), continuous or intermittent small molecule therapeutics, or any other investigational agents within a period which is ≤ 5T1/2 or ≤ 4 weeks (whichever is longer) prior to study entry
* History of somatic or psychiatric disease/condition that may interfere with the objectives and assessments of the study.
* Malignant disease, other than that being treated in this study. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within 2 years prior to study treatment; completely resected basal cell and squamous cell skin cancers; any malignancy considered to be indolent and that has never required therapy; and completely resected carcinoma in situ of any type
* pregnant or breast-feeding women
* women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, are not allowed to participate in this study UNLESS they are using highly effective methods of contraception throughout the study and for 6 months after study drug discontinuation. Highly effective contraception methods include:

  * Total abstinence
  * Male or female sterilization
  * Combination of any two of the following (a+b or a+c or b+c)

    1. Use of oral, injected, or implanted hormonal methods of contraception. In case of use of oral contraception, women should be stable on the same pill for a minimum of 3 months before taking study treatment.
    2. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
    3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository. Post-menopausal women are allowed to participate in this study. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum Follicle-Stimulating Hormone (FSH) levels > 40 mIU/mL [for US only: and estradiol < 20 pg/mL] or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to screening. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment is she considered not of child bearing potential. Sexually active males must use a condom during intercourse while taking the drug and for 6 months after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-11-27 (Actual)

PRIMARY OUTCOMES:
Phase I: Incidence of dose limiting toxicities (DLTs) of [177Lu]-NeoB | Within 42 days following the first administration of [177Lu]-NeoB
  A dose-limiting toxicity (DLT) is defined as a clinically relevant adverse event or abnormal laboratory value not attributable to the disease or disease-related processes under investigation, considered possibly related to [177Lu]-NeoB that occurs within 42 days following the first administration of [177Lu]-NeoB (cycle 1) and meets any of the criteria listed in Table 6-4 (Criteria for defining dose-limiting toxicities).
Phase I: Determination of Maximum Tolerated Dose (MTD)/ Recommended phase two dose (RP2D) of [177Lu]-NeoB | Within 42 days following the first administration of [177Lu]-NeoB
  The maximum tolerated dose (MTD) and/or the recommended phase II dose (RP2D) of [177Lu]-NeoB will be identified:
  1. MTD is defined as the lowest single dose at which 25% or more of the patients experienced a DLT during the first cycle (6 weeks).
  2. RP2D is defined as the single dose level below the MTD. The number of cycles recommended for Phase II will be defined based on the cumulative dose toxicities reported during Phase I.
Phase IIa (Cohorts A, B and C): Individual clinical responses assessed by Response Evaluation Criteria In Solid Tumors (RECIST v1.1) | 25 months
  To assess the anti-tumor activity of [177Lu]-NeoB at the RP2D across different solid tumors
Phase IIa (Cohort E): Absorbed radiation doses of [177Lu]-NeoB in organs and tumor lesions | 6 weeks
  Absorbed radiation doses in organs and tumor lesions will be summarized with descriptive statistics. Lesion number will be assigned by dosimetry expert.
Phase IIa (Cohort E): Concentration of [177Lu]-NeoB in blood over time and derived PK parameters | 6 weeks
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Concentration of [177Lu]-NeoB will be listed and summarized using descriptive statistics.
Phase I: identify maximum tolerated and/or recommended Phase II dose | 18 months
Phase II: assess disease control rate 20 weeks after completion of treatment | 18 months

SECONDARY OUTCOMES:
Phase I: Tissue Activity Curves (ACs) | 6 weeks
  Tissue activity curves (ACs) will be generated from the amount of radioactivity in one given tissue at a given moment over the amount of radioactivity present in the blood at that given moment.
Phase I: Time Activity Curves (ACs) | 6 weeks
  Time Activity Curves (ACs) describe the percentage of the activity injected versus time.
Phase I: Absorbed radiation doses of [177Lu]-NeoB in critical organs | 6 weeks
  Absorbed radiation doses in critical organs (e.g. kidneys, bone marrow, pancreas) will be summarized with descriptive statistics. Lesion number will be assigned by dosimetry expert.
Phase I: Urinary excretion of [177Lu]-NeoB | 6 weeks
  Urine samples will be collected over specified time intervals and analyzed for radioactivity using a gamma counter. The radioactivity excreted in urine will be summarized using descriptive statistics.
Phase I: Half-life of [177Lu]-NeoB in blood | 6 weeks
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. The half-live will be listed and summarized using descriptive statistics.
Phase I: Residence time of [177Lu]-NeoB in organs and tumor lesions | 6 weeks
  Residence time in organs and tumors lesions will be summarized with descriptive statistics. Lesion number will be assigned by dosimetry expert.
Phase I: Individual objective response and Duration of Response (DOR) | 25 months
  DOR is defined as the duration of time between the date of first documented response (CR or PR) in soft tissue according to PCWG3 modified RECIST 1.1, and the date of first documented progression or death due to any cause.
Phase IIa (Cohorts A, B and C): Absorbed radiation doses of [177Lu]-NeoB in organs and tumor lesions | 6 weeks
  Absorbed radiation doses in organs and tumor lesions will be summarized with descriptive statistics. Lesion number will be assigned by dosimetry expert.
Phase IIa (Cohorts A, B and C): Concentration of [177Lu]-NeoB in blood over time and derived PK parameters | 6 weeks
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Concentration of [177Lu]-NeoB will be listed and summarized using descriptive statistics.
Phase IIa (Cohorts A, B and C): Changes from baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | 15 months
  The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the patient), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the patient).
Phase IIa (Cohort E): Adverse Events for [177Lu]-NeoB when co-administered with the NEPi LCZ696 in Cycle 1 | 25 months
  The distribution of adverse events for [177Lu]-NeoB when co-administered with the neprilysin inhibitor (NEPi) LCZ696 will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.
Phase IIa (Cohort E): Dose interruptions and modifications for [177Lu]-NeoB when co-administered with the NEPi LCZ696 in Cycle 1 | Within 42 days following the first administration of [177Lu]-NeoB (Cycle 1)
Phase I and Phase IIa: Adverse Events for [177Lu]-NeoB | 25 months
  The distribution of adverse events for [177Lu]-NeoB as monotherapy will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.
Phase I and Phase IIa: Adverse Events for [68Ga]-NeoB | 25 months
  The distribution of adverse events for [68Ga]-NeoB will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.
Phase I and Phase IIa: Dose interruptions and modifications | 25 months
Determine Tissue Activity Curves (ACs) [177Lu-NeoB] | 18 months
  ratio of radioactivity in tissue vs blood
Determine Time Activity Curves | 18 months
  ratio of % activity injected vs time
Absorbed radiation dose | 18 months
  absorbed radiation dose to critical organs
Urinary excretion of [177Lu]-NeoB | 18 months
  measure amount of [177Lu]-NeoB excreted in Urine
Blood Half-life of [177Lu]-NeoB | 18 months
Organ Residence time of [177Lu]-NeoB | 18 months
Objective Response Rate | 18 months
Duration of Response | 18 months
Progression Free Survival | 18 months
Adverse Events [177Lu-NeoB] | 18 months
Dose modifications | 18 months
Adverse Events [68Ga-NeoB] | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Study Director, Study Director — Advanced Accelerator Applications
Locations (11):
- United States (6):
  - City of Hope, Duarte, California
  - Stanford University, Stanford, California
  - John Hopkins University, Baltimore, Maryland
  - Oregon Health & Science University, Portland, Oregon
  - Pittsburgh University, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Medical University of Innsbruck, Innsbruck, Austria
- CHU de Grenoble, La Tronche, France
- Erasmus MC, Rotterdam, Netherlands
- Vall d'Hebron Institute of Oncology, Barcelona, Spain
- Addenbroke's hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Taunk NK, Escorcia FE, Lewis JS, Bodei L. Radiopharmaceuticals for Cancer Diagnosis and Therapy: New Targets, New Therapies-Alpha-Emitters, Novel Targets. Cancer J. 2024 May-Jun 01;30(3):218-223. doi: 10.1097/PPO.0000000000000720. PMID 38753757
- [Derived] Sundlov A, Sjogreen-Gleisner K. Peptide Receptor Radionuclide Therapy - Prospects for Personalised Treatment. Clin Oncol (R Coll Radiol). 2021 Feb;33(2):92-97. doi: 10.1016/j.clon.2020.10.020. Epub 2020 Nov 12. PMID 33189510